CLINICAL TRIAL: NCT00287911
Title: A Phase I Study of Adjuvant Topotecan and Cisplatin With Concurrent Radiation Therapy for Advanced Cervical Cancer
Brief Title: Topotecan, Cisplatin, and Radiation Therapy in Treating Patients With Advanced Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000452043; UMN-2001LS041 (Other: CPRC, University of Minnesota); UMN-WCC-34 (Other: Women's Cancer Center, University of Minnesota); 104864/638 (Other: GlaxoSmithKline)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Topotecan; Brachytherapy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combo Chemotherapy and Radiation (Experimental): Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36. Some patients may also undergo brachytherapy. Patients also receive cisplatin intravenously (IV) over 1 hour on days 1, 8, 15, 22, 29, and 36 and topotecan IV continuously on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: cisplatin; Drug: topotecan hydrochloride; Radiation: brachytherapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — intravenously (IV) over 1 hour on days 1, 8, 15, 22, 29, and 36
  Other Names: cisplatinum; CDDP; Platinol AQ
Drug: topotecan hydrochloride — intravenously continuously on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36 -Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined
  Other Names: Hycamtin
Radiation: brachytherapy — Some patients may also undergo brachytherapy
Radiation: radiation therapy — once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36
  Other Names: radiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Topotecan and cisplatin may make tumor cells more sensitive to radiation therapy. Giving topotecan and cisplatin together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of topotecan when given together with cisplatin and radiation therapy in treating patients with advanced cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of topotecan when administered with cisplatin in patients with advanced cervical cancer.
* Identify any unique toxicities associated with administering radiotherapy along with adjuvant cisplatin and topotecan in patients with cervical cancer.
* Determine the feasibility of administering continuous infusion topotecan chemotherapy together with radiation therapy.
* Assess the quality of life of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of topotecan.

Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36. Some patients may also undergo brachytherapy. Patients also receive cisplatin intravenously (IV) over 1 hour on days 1, 8, 15, 22, 29, and 36 and topotecan IV continuously on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Quality of life is assessed at baseline and at 4 and 14 weeks after completion of study treatment.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical carcinoma

  * Deemed not curable by surgery or radiotherapy alone
  * The following stages are eligible:

    * Stage IIB
    * Stage IIIA or IIIB
    * Stage IVA
    * Stage IB or IIA with ≥ 1 of the following risk factors:

      * Primary tumor ≥ 6 cm
      * Positive pelvic and/or para-aortic lymph nodes (resected or unresected)
      * Positive surgical margins
      * Depth of invasion > 50% and positive capillary-lymphatic space involvement
* The following histologic subtypes are eligible:

  * Squamous
  * Adenosquamous
  * Adenocarcinoma
* No recurrent cervical cancer
* Gynecologic Oncology Group (GOG) performance status 0, 1, or 2
* White blood cells (WBC) ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Granulocyte count ≥ 1,500/mm^3
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 1.5 times institutional normal
* Serum glutamic oxaloacetic transaminase (SGOT) and alkaline phosphatase ≤ 3 times institutional normal
* No other prior or concurrent malignancies other than skin (excluding melanoma)
* No septicemia, severe infection, gastrointestinal bleeding, or intestinal obstruction
* No anatomic abnormalities (e.g., pelvic kidney or renal transplant) requiring modification of radiation fields
* Fertile patients must use effective contraception
* Negative pregnancy test
* Patients with evidence of abnormal cardiac conduction (e.g., bundle branch block, heart block) are eligible if disease is stable for the past 6 months
* Recovered from recent surgery

Exclusion Criteria:

* Prior pelvic radiation
* Pregnant or nursing
* History of thrombus
* History of unstable angina or myocardial infarction within the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of topotecan | Week 3 After First Course of Therapy
  Adequate Response Trial Minimum length of trial to evaluate response is defined as receiving the first course of chemotherapy and living at least three weeks for repeat measurement to be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Linda F. Carson, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States